CLINICAL TRIAL: NCT05400343
Title: Efficacy of Lung and Inferior Vena Cava Sonography for Fluid Optimization in Critically Ill Patients With Traumatic Brain Injury
Brief Title: Efficacy of Lung and Inferior Vena Cava Sonography for Fluid Optimization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: MFM-IRB, MD ∕ 22.01.591
Record Dates: First submitted 2022-05-27; First posted 2022-06-01 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Standard of Care; Control Groups

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single-blind (participant) study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (control group) (Active Comparator): fluid therapy will be guided by conventional ICU policies to maintain an adequate intravascular volume and good urine output
  Interventions: Procedure: Standard care (control group); Other: Standard ICU Care
- US-guided ﬂuid management (active group) (Experimental): Fluid therapy will be guided by measurements of lung and IVC sonography
  Interventions: Procedure: US-guided ﬂuid management (active group); Other: Standard ICU Care

INTERVENTIONS:
Procedure: Standard care (control group) — Following 24 hours from admission to the ICU, the standard care will be continued according to conventional ICU protocols
  The mean fluid intake will range from (2-3L per day) targeting zero or slightly negative balance (up to - 300ml). Various parameters will be used to attain this goal based on case-by-case clinical judgment.
  Arms: Standard care (control group)
Procedure: US-guided ﬂuid management (active group) — Within 24 hours from admission to the ICU, IVC and lung sonography will be performed every other day and according to their measurements, the volume of fluid therapy will be adjusted.
  Arms: US-guided ﬂuid management (active group)
Other: Standard ICU Care — All patients will receive the usual care for 24 hours according to ICU policies. The main target is to maintain an adequate intravascular volume and good urine output. The mean fluid intake will range from (2-3L per day) targeting zero or slightly negative balance (up to - 300ml). Various parameters will be used to attain this goal based on case-by-case clinical judgment. Lung sounds, heart rate, blood pressure, temperature, urine output, Lactate, haemoglobin, haematocrit, serum urea, creatinine, sodium, potassium, chloride, and bicarbonate values

SUMMARY:
Traumatic brain injury (TBI) is a leading cause of death and disability in trauma patients. As the primary injury cannot be reversed, management strategies must focus on preventing secondary injury by avoiding hypotension and hypoxia and maintaining appropriate cerebral perfusion pressure (CPP), which is a surrogate for cerebral blood flow (CBF). The goal should be euvolemia and avoidance of hypotension. The assessment of a patient's body fluid status is a challenging task for modern clinicians.

The use of Ultrasonography to assess body fluids has numerous advantages. The concept of using lung ultrasound for monitoring the patient is one of the major innovations that emerged from recent studies. Pulmonary congestion may be semiquantiﬁed using lung ultrasound and deciding how the patient tolerates fluid. Inferior vena cava (IVC) sonography and point-of-care ultrasound (POCUS) has become widely used as a tool to help clinicians prescribe ﬂuid therapy. Common POCUS applications that serve as guides to ﬂuid administration rely on assessments of the inferior vena cava to estimate preload and lung ultrasound to identify the early presence of extravascular lung water and avoid ﬂuid over resuscitation In this study we will use the measurements of both lung and IVC together to guide fluid dosage in critically ill patients with TBI. We will also use ONSD as a mirror for intra-cranial pressure (ICP).

DETAILED DESCRIPTION:
The aim of this study is to detect the effectiveness of using IVC and lung ultrasound as bedside tools to ensure euvolemia in patients with traumatic brain injuries

Positive fluid balances have been associated with (angiographic) vasospasm, longer hospital length of stay and poor functional outcomes The assessment of a patient's body fluid status is a challenging task for modern clinicians. Currently, the most accurate method to guide ﬂuid administration decisions uses "dynamic" measures that estimate the change in cardiac output that would occur in response to a ﬂuid bolus. Unfortunately, their use remains limited due to required technical expertise, costly equipment, or applicability in only a subset of patients. Alternatively, point-of-care ultrasound (POCUS) has become widely used as a tool to help clinicians prescribe ﬂuid therapy.

International recommendations suggest that the inferior vena cava (IVC) can be assessed to estimate the pressure in the right atrium of non-ventilated patients because of its collapsibility during inspiration. An IVC diameter of < 21mm with collapsibility of > 50% during inspiration suggests normal right atrium pressure (between 0 and 5 mmHg), whereas a diameter of > 21mm with collapsibility of < 50% suggests high pressure (between 10 and 20mmHg). The dynamic method of IVC evaluation, based on the variation in its diameter with respiration, enables the assessment of the potential benefit of fluid administration as a function of IVC compliance.

Ultrasonography of optic nerve sheath diameter (ONSD) in TBI patients has been shown to correlate with increased ICP and systemic reviews have supported this observation.

In this study, we will use the measurements of both lung and IVC together to guide fluid dosage in critically ill patients with TBI. We will also use ONSD as a mirror for ICP

The study investigates the effect of using bedside sonography in fluid assessment in a critically ill patient

ELIGIBILITY:
Inclusion Criteria:

* BMI less than 35 kg/m2
* Diagnosed with traumatic brain injury
* Glasgow coma score ≥ 4

Exclusion Criteria:

* Inability to get consent
* Presence of Increased intra-abdominal pressure,
* Presence of acute cor pulmonale
* Presence of severe right ventricular dysfunction.
* Pregnancy
* Patients with known pulmonary conditions that interfere with the interpretation of lung ultrasound like pneumectomy; pulmonary fibrosis; persistent pleural effusion
* Stage 5 chronic kidney disease
* indication for emergency renal replacement therapy (RRT)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-06-15 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Cumulative Fluid balance | 10 days or until ICU discharge which comes first.
  The difference between patient fluid intake and patient fluid output is recorded every 24 h then the cumulative balance is recorded

SECONDARY OUTCOMES:
ONSD as mirror for intracranial pressure. | every other day for 10 days or until ICU discharge which comes first
  Ultrasonic examination will be performed by an experienced investigator with a 11-3 MHz linear transducer. The patients will be examined in a supine position with the head elevated at 20-30° ONSD was defined as the distance between the external borders of the hyperechoic area 3 mm posterior to the point where the optic nerve entered the globe, using an electronic caliper along the axis perpendicular to the retina. . To minimize intraobserver variability, each measurement was performed three times and the mean value was derived
Urine output | 10 days or until ICU discharge which comes first
  patient urine output per ml is collected and recorded every 6 hours and total daily urine output is recorded
Frequency of hypotension | every other day for 10 days or until ICU discharge which comes first
  hypotension is defined as systolic blood pressure less than 90 mmHg, or diastolic blood pressure less than 50 mmHg or both or more than 20 % decline in basal blood pressure for more than 5 minutes.
Duration of hypotension | 10 days or until ICU discharge which comes first
  every other day for 10 days or until ICU discharge which comes first
Serum creatinine | 10 days or until ICU discharge which comes first
  daily serum creatinine in mg /dl is ordered and recorded
Incidence of pulmonary edema | 10 days or until ICU discharge which comes first
  Diagnosis of the patient with pulmonary edema by (x ray, CT, pulse oximetry, other methods) is recorded
Length of mechanical ventilation | 10 days or until ICU discharge which comes first
  Duration of mechanical ventilation in days is record
Mortality at 10 days | mortality at day 10

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa M Saied, MD, Study Chair — Professor of Anesthesia and Surgical Intensive Care; Medhat M Messeha, MD, Study Director — Assistant Professor of Anesthesia and Surgical Intensive Care
Locations (1):
- Mansoura University, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant individual data for all primary and secondary outcomes will be made available
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 6 months of study completion Data will be available for audits and quantitative meta-analyses for 10 years
Access Criteria: Data access requests will be reviewed by an external independent review panel. Requestors will be required to sign a Data Access Agreement